CLINICAL TRIAL: NCT00795496
Title: Bronchial Hyperreactivity in Atopic Dermatitis Patients - a 10 Year Follow-up
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Sakari Reitamo, MD, PhD, Specialist in Dermatology, Acting Professor, Helsinki University Central Hospital, Department of Dermatology
Other Study IDs: 232685
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2008-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Bronchial hyperreactivity; Skin prick tests; Serum IgE; Mantoux test
MeSH Terms: conditions — Dermatitis, Atopic; Bronchial Hyperreactivity

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — Serum is collected for measurement of IgE
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AD patients: AD patients who fulfill the inclusion criteria for the study
  Interventions: Procedure: Histamine provocation; Procedure: Skin prick tests; Procedure: Serum IgE blood testing; Procedure: Mantoux-testing

INTERVENTIONS:
Procedure: Histamine provocation — A dosimetric histamine challenge test in which the provocative dose of inhaled histamine producing a decrease of 15% in FEV1 is measured.
Procedure: Skin prick tests — Skin prick testing will be performed for: birch, timothy, mugwort, alder, pine, cat, dog, horse, house dust mite, Cladosporium herbarum.
Procedure: Serum IgE blood testing — One blood test to measure total serum IgE
Procedure: Mantoux-testing — Tuberculin (2 TU) s.c. on the forearm. The test is read after 72 hours.

SUMMARY:
The investigators will contact 64 patients with atopic dermatitis (AD) who participated in a long-term tacrolimus ointment trial in Helsinki 10 years ago, and ask them to participate in this follow-up study. The investigators will do the same tests as 10 years ago, i.e. bronchial hyperreactivity, skin prick tests, serum-IgE, Mantoux-test (2 TU), and questionnaires about asthma and allergic rhinitis symptoms. The investigators also collect data about their AD medication during the last 10 years.

The investigators hypothesis is that when the skin condition improves in patients with AD the brochial hyperreactivity improves. The investigators also want to study whether different treatments play a role in the development or resolution of bronchial hyperreactivity.

DETAILED DESCRIPTION:
We will by letters and telephone contact all patients (n=64) who fulfill the inclusion criteria for this study.

The testing in the study (bronchial hyperreactivity, skin prick testing, serum IgE) is cross-sectional, but we retrospectively collect data from the last 10 years about the skin condition and medication for atopic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patient has participated in the FG-506-06-21 study in Helsinki
* Patient was tested for bronchial hyperreactivity in the years 1998-2000
* Patient gives signed informed consent to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators invite all patients who participated in the FG-506-06-21 tacrolimus ointment study, and who at baseline in that study were tested for bronchial hyperreactivity.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Bronchial hyperreactivity | 10 year follow-up

SECONDARY OUTCOMES:
Skin prick tests | 10 year follow-up
Serum-IgE | 10-year follow-up
Mantoux-test | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sakari Reitamo, MD, PhD, Principal Investigator — Skin- and Allergy Hospital, Dep. of Dermatology
Locations (1):
- Skin- and Allergy Hospital, Department of Dermatology, Helsinki, Finland

REFERENCES:
- [Background] Virtanen H, Remitz A, Malmberg P, Rytila P, Metso T, Haahtela T, Reitamo S. Topical tacrolimus in the treatment of atopic dermatitis--does it benefit the airways? A 4-year open follow-up. J Allergy Clin Immunol. 2007 Dec;120(6):1464-6. doi: 10.1016/j.jaci.2007.08.021. Epub 2007 Oct 1. No abstract available. PMID 17910892